CLINICAL TRIAL: NCT03488875
Title: The Impact of Mindfulness-Based Resilience Training on Stress-Related Biological, Behavioral, and Health-Related Outcomes in Law Enforcement Officers
Brief Title: Impact of Mindfulness Training on Stress-related Health Outcomes in Law Enforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1529; 2017-R2-CX-0033 (Other Grant/Funding Number: National Institute of Justice); A483000 (Other: UW, Madison); L&S (Other: UW, Madison)
Record Dates: First submitted 2018-03-22; First posted 2018-04-05 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Stress, Psychological; Sleep; Inflammation; Mental Health
MeSH Terms: conditions — Stress, Psychological; Inflammation; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants are randomized to an active treatment group and a waitlist control group.
Masking Description: Participants cannot be made blind to study assignment due to the nature of the intervention.
  Baseline (T1) measures will be collected prior to treatment assignment. Every effort will be taken to minimize knowledge of group assignment by the study team, in particular the PI and other individuals involved in data analysis; however, the small size of the study team and overlapping roles of team members may preclude masking of group assignment for all members of the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mMBRT (Experimental): Individuals in the mMBRT group will receive an 8-week mindfulness-based intervention in groups of approximately 15 individuals in 8 weekly 2-hour classes (one of these classes, toward the end of the course, is approximately 4 hours and integrates many of the practices and teachings covered throughout the training program).
  Interventions: Behavioral: mMBRT
- Waitlist control group (No Intervention): Individuals in the waitlist control group will complete the same assessments as those in the active treatment group, but will not be offered any intervention until the conclusion of the trial. At this time, control group participants will be offered the intervention.

INTERVENTIONS:
Behavioral: mMBRT — Madison Mindfulness-Based Resilience Training (mMBRT) is an 8-week mindfulness-based intervention developed specifically for police officers, which is similar to and inspired by a program developed by researchers at Pacific (OR) University (Christopher, Goerling et al., 2016). mMBRT includes 8 weekly 2-hour classes involving guided meditation practice, gentle movement, and group-based discussion (the 7th class is a longer, 4-hour class). The total class time is about 18 hours over 8 weeks, and participants are asked to engage in home practice for up to 30 minutes/day, 6 days/week throughout the intervention.
  Other Names: Madison Mindfulness-Based Resilience Training; MBRT
  Arms: mMBRT

SUMMARY:
In a sample of 120 officers from Dane County law enforcement agencies, the investigators are conducting a randomized controlled trial of an 8-week mindfulness-based training program for police officers, Madison Mindfulness-Based Resilience Training (mMBRT), and investigating the impact of this training on subjective responses to stress, stress-related psychological and physical health outcomes, and biological and behavioral correlates of perceived stress. While the benefits of mindfulness-based interventions have been documented in a variety of populations, this will be the largest and most comprehensive study of its kind of law enforcement personnel. In addition to self-report measures, this study assesses an array of objective biological and behavioral outcomes both in the laboratory and in the field that may speak to mechanisms of change involved in symptom reduction.

DETAILED DESCRIPTION:
120 police officers will be recruited from Dane County law enforcement agencies to take part in an 8-week, group-based, mindfulness-based training program called Madison Mindfulness-Based Resilience Training (mMBRT). Officers will be randomized to an active group, which will receive mMBRT immediately after baseline assessments, and a waitlist control group, which will receive mMBRT after a post-intervention assessment and a subsequent follow-up assessment. mMBRT is similar to and inspired by MBRT, and both of these programs are law enforcement-specific interventions based on Mindfulness-Based Stress Reduction (MBSR), a commonly used mindfulness program in many healthcare settings. mMBRT is structurally similar to MBSR, with 8 weekly 2-hour classes involving guided meditation practices, gentle movement, and group-based discussion (one of these classes, toward the end of the course, is approximately 4 hours and integrates many of the practices and teachings covered throughout the training program). Participants will be provided with weekly homework assignments and audio recordings that provide guided instruction in various meditation and yoga practices.

At three separate timepoints, officers will take part in a laboratory assessment that involves the following procedures:

* administration of computerized behavioral tasks
* completion of self-report questionnaires that assess trauma history and occupational stressors, perceived stress, sleep, physical and mental health
* collection of a small amount of blood via finger prick and/or venipuncture (to assess peripheral inflammatory markers)
* collection of a small amount of hair from the scalp (to assess hair cortisol concentration)
* measurement of height and weight for the assessment of body mass index, and for use with activity trackers data

In conjunction with these laboratory assessments, data will be collected from officers in the field over the course of approximately 1 week (coinciding with a regularly scheduled work week), including the following procedures:

* officers will wear an activity monitor (e.g., Fitbit) to allow for objective monitoring of sleep quality and resting heart rate throughout the study
* officers will collect saliva samples 4 times per day over 3 days for the assessment of salivary cortisol
* officers will complete daily logs of work hours, types of events encountered during work, perceived stress related to these events, and self-reported mood and affect ratings

These field data will be related to dispatch records, which will provide objective information regarding the types of incidents responded to, and the time and location of these incidents.

The laboratory and field assessments will be collected at baseline (prior to randomization); after the active mMBRT group completes the intervention; and at a follow-up visit (approximately 4 months after the end of the intervention), after which the wait-list group will be offered the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Capable of giving informed consent
* Fluent in English
* Currently employed sworn law enforcement officer working in the Dane County Sheriff's Office, Madison Police Department, or University of Wisconsin-Madison Police Department.

Exclusion Criteria:

* Extensive prior experience in meditation practice, or previous completion of Mindfulness-Based Stress Reduction, Mindfulness-Based Resilience Training, or a substantively similar meditation training program
* A work schedule that precludes one from committing to regular participation in the 8-week training program
* Command staff working in a supervisory role

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Change in perceived occupational stress | Baseline, post-intervention (3 months)
  Change in combined scores of perceived operational and organizational stressors from the Police Stress Questionnaire (McCreary & Thompson, 2004) from baseline to 3 months. Each of these 2 scales has 20 items with 1-7 ratings, where higher scores indicate greater stress (1=no stress at all, 7=A lot of stress). Organizational and operational stress scales will be summed to create a single value with a range of 40-280.
Change in diurnal cortisol slope | Baseline, post-intervention (3 months)
  Saliva samples collected on each of 3 days will be used to calculate diurnal cortisol slope, defined as the change between the peak cortisol response in the 45 minutes after awakening and cortisol levels just prior to bedtime, with a hypothesized steeper slope in the intervention vs. waitlist group at post-intervention (3 months) vs. baseline.

SECONDARY OUTCOMES:
Change in cortisol awakening response | Baseline, post-intervention (3 months)
  The cortisol awakening response (CAR) will be measured using saliva samples collected 0, 30, and 45 minutes after awakening on each of 3 days, with hypothesized increased CAR in the intervention vs. waitlist group at post-intervention (3 months) vs. baseline.
Change in peripheral inflammatory markers | Baseline, post-intervention (3 months)
  Composite of hsCRP and 4-plex of pro-inflammatory cytokines (IL-6, IL-8, IL-10, TNF-alpha) is hypothesized to be lower in intervention vs. waitlist group at post-intervention (3 months) vs. baseline.
Change in hyperarousal symptoms | Baseline, post-intervention (3 months), follow-up (6 months)
  Change in hyperarousal symptoms from the PTSD Checklist for DSM-5 at post-intervention (3 months) vs. baseline
Change in subjective sleep quality | Baseline, post-intervention (3 months)
  Global scores on the Pittsburgh Sleep Quality Index (Buysse et al., 1988) will be compared at post-intervention (3 months) vs. baseline
Change in perceived stress | Baseline, post-intervention (3 months)
  Changes in total scores from the Perceived Stress Scale (10-item version; Cohen et al., 1988) from baseline to 3 months.

OTHER OUTCOMES:
Change in hair cortisol concentration | Baseline, follow-up (6 months)
  Hair cortisol concentration will be assessed from a 3-cm sample of hair collected from participants' scalps, corresponding to approximately 3 months of hair growth, at 6 months vs. baseline.
Change in restful minutes of sleep | 5-7 nights of sleep will be monitored at baseline and post-intervention (3 months)
  Change in minutes of behaviorally assessed restful sleep time during 1 week of sleep measured in the field using Fitbit Charge 2 activity trackers at post-intervention (3 months) vs. baseline.
Change in behavioral pattern separation ability | Baseline, post-intervention (3 months)
  Changes in lure discrimination index (LDI) scores from the Mnemonic Similarity Task (Stark et al., 2015) will be assessed between baseline and post-intervention (3 months). LDI scores have a theoretical range of -1 to +1, where a score of +1 indicates perfect ability to discriminate novel items from those previously seen and 0 indicates chance discrimination of novel from previously seen items. Negative scores, while theoretically possible, are rare as they indicate greater labeling of novel items as "old" compared to previously seen items as "old".'
Change in mood and anxiety symptoms | Baseline, post-intervention (3 months)
  Change in depression and anxiety subscale scores from the 43-item version of the Patient-Reported Outcomes Measurement Information System (PROMIS-43) at post-intervention (3 months) vs. baseline. There are 6 depression and 6 anxiety items, each of which is scored on a scale of 1 ("never") to 5 ("always"), yielding a range of 6-30 for each subscale with higher scores indicating greater impairment.
Change in total PTSD symptoms | Baseline, post-intervention (3 months)
  Change in total PTSD symptoms from the PTSD Checklist for DSM-5 at post-intervention (3 months) vs. baseline
Change in resting heart rate | Baseline, post-intervention (3 months)
  Changes in average resting heart rate calculated over 3-7 days of field data collection using a Fitbit Charge 2 activity tracker at post-intervention (3 months) vs. baseline.
Change in pain interference | Baseline, post-intervention (3 months)
  Change in pain interference subscale scores from the 43-item version of the Patient-Reported Outcomes Measurement Information System (PROMIS-43) at post-intervention (3 months) vs. baseline.
Change in burnout | Baseline, post-intervention (3 months)
  Change in the two core dimensions of burnout, exhaustion and disengagement, on the Oldenburg Burnout Inventory (Halbesleben & Demerouti, 2005) at post-intervention (3 months) vs. baseline.
Change in work productivity | Baseline, post-intervention (3 months)
  Change in work productivity, measured as the estimated percentage of work time affected by chronic mental and physical health issues on the Work Limitations Questionnaire (short form; Lerner et al., 2001) at post-intervention (3 months) vs. baseline.
Change in good health practices | Baseline, post-intervention (3 months)
  Change in physical health and well-being behaviors as measured by the Good Health Practices Scale (Hampson et al., 2017) at post-intervention (3 months) vs. baseline.
Change in self-reported mindfulness | Baseline, post-intervention (3 months)
  Changes in total scores and individual dimensions of the Five-Facet Mindfulness Scale (short form; Bohlmeijer et al., 2011) at post-intervention (3 months) vs. baseline.
Change in work-family spillover | Baseline, post-intervention (3 months)
  Change in work-to-family and family-to-work spillover from the Work-Family Spillover Scale (Grzywacz & Marks, 2000) at post-intervention (3 months) vs. baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Grupe, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Center for Healthy Minds, University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Grupe DW, Stoller JL, Alonso C, McGehee C, Smith C, Mumford JA, Rosenkranz MA, Davidson RJ. The Impact of Mindfulness Training on Police Officer Stress, Mental Health, and Salivary Cortisol Levels. Front Psychol. 2021 Sep 3;12:720753. doi: 10.3389/fpsyg.2021.720753. eCollection 2021. PMID 34539521
- [Derived] Chen S, Grupe DW. Trait Mindfulness Moderates the Association Between Stressor Exposure and Perceived Stress in Law Enforcement Officers. Mindfulness (N Y). 2021;12(9):2325-2338. doi: 10.1007/s12671-021-01707-4. Epub 2021 Aug 5. PMID 34377216